CLINICAL TRIAL: NCT03303781
Title: BeSingCardioRehab: An Intercontinental Retrospective Cohort Study Comparing Cardiac Rehabilitation in Belgium and Singapore
Brief Title: BeSingCardioRehab: CR in Belgium Versus Singapore
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, prof. dr., Hasselt University
Other Study IDs: BeSingCardioRehab01
Record Dates: First submitted 2017-09-28; First posted 2017-10-06 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- BE + CR: Belgian ischemic heart disease patients with cardiac rehabilitation program
  Interventions: Other: Cardiac Rehabilitation
- BE-CR: Belgian ischemic heart disease patients without cardiac rehabilitation program
- Si + CR: Singapore (Asian) ischemic heart disease patients with cardiac rehabilitation program
  Interventions: Other: Cardiac Rehabilitation
- SI -CR: Singapore (Asian) ischemic heart disease patients without cardiac rehabilitation program

INTERVENTIONS:
Other: Cardiac Rehabilitation — phase II center-based cardiac rehabilitation
  Groups: BE + CR; Si + CR

SUMMARY:
Background: Cardiac rehabilitation is indicated for ischemic heart disease patients; the program content of which is well described in both European and American guidelines. In contrast, literature on cardiac rehabilitation program content and efficacy in the Asian population is sparse.

Methods: BeSingCardioRehab will be an intercontinental, retrospective cohort study conducted in two cardiac rehabilitation referral centers in Belgium and Singapore. The first aim is to compare the impact of phase II center-based cardiac rehabilitation on Major Adverse Cardiac Events for ischemic heart disease patients between Europe (i.e. Belgian) and Asia (i.e. Singaporean) in the long-term. The second objective is to compare the efficacy of phase II cardiac rehabilitation on short-term morbidity (assessed with the validated SMART Risk Score) between index European and Asian ischemic heart disease patients. The level of compliance of the Belgian and Singaporean cardiac rehabilitation programs to European guidelines standards will also be evaluated.

Hypotheses BeSingCardiorehab will be one of the first studies assessing cardiac rehabilitation in Asia. Based on the BeSingCardioRehab study results, phase II center-based cardiac rehabilitation programs, can/will be adapted in order to improve program content and outcomes.

DETAILED DESCRIPTION:
BeSingCardioRehab is an intercontinental, multi-center, retrospective cohort study conducted in two cardiac rehabilitation referral centers (Heart Center Hasselt in Belgium and National Heart Center Singapore in Singapore).

Patients will be divided in four groups (1:1:1:1) based on i. whether or not they received phase II cardiac rehabilitation and ii. whether they are from Belgium or Singapore.

The first objective of BeSingCardioRehab is to compare the impact of phase II center-based cardiac rehabilitation on Major Adverse Cardiac Events for ischemic heart disease patients between Europe (i.e. Belgian) and Asia (i.e. Singaporean) in the long-term. The second objective is to compare the efficacy of phase II cardiac rehabilitation on short-term morbidity (assessed with the validated SMART Risk Score) between index European and Asian ischemic heart disease patients. The level of compliance of the Belgian and Singaporean cardiac rehabilitation programs to European guidelines standards will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

i. patients in the revascularised, stabilized and asymptomatic phase following an acute coronary syndrome (ACS) (unstable angina, non ST-elevation ACS or ST-elevation ACS)

ii. patients initially presenting with stable angina who are revascularised or asymptomatic under optimal medical treatment (not amenable for revascularization).

Exclusion Criteria:

i. end-stage chronic kidney disease (stage V, GFR < 15 ml/min/1.73 m2 and/or dialysis) ii. severe chronic obstructive pulmonary disease (COPD) (GOLD stage III-IV, Tiffeneau index < 0.70 and FEV1 < 49% of normal) iii. terminal cancer with a prognosis of < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ligible study participants include patients suffering from stable ischemic heart disease, enrolled in phase II center-based cardiac rehabilitation. Stable ischemic heart disease is defined as i. patients in the revascularised, stabilized and asymptomatic phase following an acute coronary syndrome (ACS) (unstable angina, non ST-elevation ACS or ST-elevation ACS) or ii. patients initially presenting with stable angina who are revascularised or asymptomatic under optimal medical treatment (not amenable for revascularization) [2-4]. Phase II cardiac rehabilitation is defined as the secondary prevention center-based intervention performed following the index cardiovascular disease event with the aim of clinical stabilization, risk stratification, and promotion of a long-term healthy status.
Sampling Method: Probability Sample
Enrollment: 2792 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
MACE | From date of index hospitalisation to a common stopping date (1 September 2017).
  The primary endpoint is MACE, which is a composite of death from cardiovascular causes, non-fatal myocardial infarction, or non-fatal stroke [13] in the long-term.

SECONDARY OUTCOMES:
SMART Risk Score | week 12
  The secondary endpoint is the short-term cardiovascular risk, assessed by the validated SMART Risk Score. Short-term is defined as 12 weeks after the index ischemic heart disease event.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dendale, Principal Investigator — Jessa Hospital
Locations (2):
- Jessa Hospital, Hasselt, Belgium
- National Heart Center Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided